CLINICAL TRIAL: NCT06339203
Title: Wound Irrigation With Saline Versus Hypodilute-chlorhexidine After Cesarean Section: a Randomized Clinical Trial (WISHES Study)
Brief Title: Wound Irrigation With Saline Versus Hypodilute-chlorhexidine After Cesarean Section (WISHES Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: Irrimax Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5240002
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Cesarean Section Complications; Cesarean Section; Infection
MeSH Terms: conditions — Infections | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Irrisept (Experimental): The experimental arm will receive irrigation solution Irrisept administered through a proprietary bottle (jet lavage) following the closure of the fascia in Cesarean section.
  Interventions: Device: Irrisept
- Normal Saline (Active Comparator): The active comparator arm will receive the standard of care irrigation solution, normal saline, administered via standard pour over following the closure of the fascia in Cesarean section.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Device: Irrisept — 450ml low concentration (0.05%) Chlorhexidine Gluconate (CHG) in 99.95% Sterile Water
  Arms: Irrisept
Drug: Normal Saline — 450mL
  Arms: Normal Saline

SUMMARY:
This investigator-initiated, open-label, randomized controlled trial will explore the effects of two treatment arms, comparing standard treatment with normal saline against Irrisept, a jet lavage solution containing a low concentration of Chlorhexidine Gluconate (CHG) at 0.05% in 99.95% sterile water for irrigation. The study aims to evaluate the impact on postoperative wound healing in patients who have undergone cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Singleton pregnancy
* Planned cesarean delivery at gestational age 37 weeks or later at Loma Linda University Children's Hospital
* Planned post-operative follow up with Loma Linda OBGYN
* Speak English or Spanish
* At least one of the following medical complications: Obesity BMI>= 30kg/m2, Diabetes, Spontaneous rupture of membranes, Intraamniotic infection

Exclusion Criteria:

* Emergency cesarean delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 400 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Composite wound evaluation scale after caesarean delivery | Up to 8 weeks postop
  Wound Evaluation scale will be used to evaluate appropriate healing in the following categories: redness, bruising, discharge, tissue breakdown, wound infection

CONTACTS AND LOCATIONS:
Overall Officials: Ruofan Yao, MD, MPH, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No